CLINICAL TRIAL: NCT02660255
Title: Safety and Tolerability of Cannabidiol in Subjects With Drug Resistant Epilepsy
Acronym: CBD
Status: Approved for marketing | Type: Expanded Access
Sponsor: University of Nebraska (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 0719-15-FB
Record Dates: First submitted 2015-12-21; First posted 2016-01-21 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Epilepsy
Keywords: CBD; Epidiolex; Myoclonic; Brain Disease; Central Nervous System Disease; GWP42003
MeSH Terms: conditions — Epilepsy; Brain Diseases; Central Nervous System Diseases | interventions — Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — Formulation: 100mg/ml CBD (Epidiolex) Solution
  Other Names: Epidiolex

SUMMARY:
This is an observational, open-label, flexible dose study that will prospectively and longitudinally assess the effect of Cannabidiol (CBD) therapy in patients with drug-resistant epilepsies through a Physician Expanded Access Investigational New Drug protocol.

DETAILED DESCRIPTION:
This study will test if Cannabidiol (CBD) therapy is safe in humans and reduces the number and/or severity of seizures in patients with drug resistant epilepsy when taken in addition to current anti-epileptic drugs (AEDs).

To be eligible, subjects must:

* have drug-resistant epilepsy
* be between 1 and 60 years of age

Subjects may participate for up to 2 years and may continue to receive the drug as available, until the compassionate use is terminated or the drug becomes approved by the FDA.

The study includes:

* Baseline, Screening and 2 phone calls
* 12 week drug titration (6 visits) and 5 phone calls
* Approximately 1 year and 9 month Treatment period (7 visits)

Subjects will come in for visits approximately every two weeks for the first three months and then quarterly for the remainder of the study. Subjects' antiepileptic drug levels will be tested to monitor for drug interactions. Lab assessments (complete blood count,CBC; comprehensive metabolic panel, CMP; urinalysis) will be performed to monitor for changes in bone marrow, liver, and kidney function to ensure safe use.

Cannabidiol will be in the form of 100 mg/ml oral solution. Subjects will be given CBD to take in addition to their current anti-epileptic drug (AED) regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 1-60 years of age.
2. Patient must have at least 4 clinically countable seizures per month. They must also have prior concomitant video-EEG with evidence documenting a diagnosis of epilepsy. Seizure history to include a documented history of generalized seizures (drop attacks, atonic, tonic-clonic and/or myoclonic), focal seizures without loss of consciousness with a motor component, focal seizures with loss of consciousness, or focal seizures with secondary generalization.
3. Drug resistant epilepsy defined as a trial of at least four drugs, including one trial of a combination of two concomitant drugs, without successful seizure control. Vagal nerve stimulation, responsive neurostimulation, RNS, deep brain stimulation, or the ketogenic diet can be considered equivalent to a drug trial and documented evidence of drug and other therapeutic failures.
4. Between 1-4 baseline anti-epileptic drugs at time of enrollment. Vagus nerve stimulator (VNS), ketogenic diet and modified Atkins diet do not count toward this limit and are not contraindicated for inclusion.
5. Subject and family sign assent (if capable)/consent/research authorization and are able to meet the study expectations for appointments for the duration of the study
6. VNS, if in use must be on stable settings for a minimum of 1 month.
7. If on ketogenic diet, must be on stable ratio for a minimum of 3 months.
8. Patients or their caregivers must be able to consistently maintain a seizure diary for at least 2 months prior to enrollment and during the course of the study period.
9. Must be Nebraska state resident.

Exclusion Criteria:

1. Renal, hepatic, pancreatic, or hematologic dysfunction as evidenced by: values above upper limits of normal for blood urea nitrogen (BUN)/creatinine, or values twice the upper limit of normal for serum transaminases [alanine transaminase (ALT), serum glutamic pyruvic transaminase (SGPT), aspartate transaminase (AST), serum glutamic-oxaloacetic transaminase (SGOT)], values twice the upper limit of normal for serum lipase and amylase, platelets <80,000 /miroliter (mcL), white blood cell count (WBC)<3.0 103 /mcL
2. Less than 4 countable (non-countable seizures includes absence and myoclonic) seizures per month
3. Use of cannabis-related product within last 30 days
4. Active substance abuse/addiction.
5. CBD is contraindicated in pregnancy and breastfeeding. Female subjects who are pregnant will be excluded from the study. If a female subject is able to become pregnant, she will be given a urine pregnancy test before entry into the study. Female subjects will be informed not to become pregnant while taking cannabidiol, and must agree to an acceptable method of barrier contraception use during the study which should include abstinence or a double barrier method for the duration of treatment.

   Female subjects must tell the investigator and consult an obstetrician or maternal-fetal specialist if they become pregnant during the study. If pregnancy occurs, CBD will be stopped in the most clinically appropriate manner.
6. Allergy to CBD or any cannabinoid.
7. Unable to provide consent and no Legally Authorized Representative (LAR) available
8. Unable to comply with study visits/requirements.
9. Use of alcohol

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Madhavan, MD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States